CLINICAL TRIAL: NCT06835972
Title: A Phase 1b/2 Study of Abemaciclib Plus Cabozantinib in Immune Checkpoint Blockade-pretreated Metastatic Clear Cell Renal Cell Carcinoma
Brief Title: A Study of Abemaciclib and Cabozantinib in People With Clear Cell Renal Cell Carcinoma (ccRCC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry); Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-126
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Renal Cell Carcinoma; Translocation Renal Cell Carcinoma
Keywords: Abemaciclib; Cabozantinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — abemaciclib; cabozantinib

STUDY DESIGN:
Intervention Model Description: This is a two-site single-arm open-label phase 1b/2 clinical trial evaluating abemaciclib plus cabozantinib in patients with metastatic ccRCC and tRCC that have progressed on therapy. The study comprises a dose escalation portion followed by a dose expansion phase 2 trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abemaciclib and Cabozantinib (Experimental): This is a two-site single-arm open-label phase 1b/2 clinical trial evaluating abemaciclib plus cabozantinib in patients with metastatic ccRCC and tRCC that have progressed on therapy. The study comprises a dose escalation portion followed by a dose expansion phase 2 trial.
  Interventions: Drug: Abemaciclib; Drug: Cabozantinib

INTERVENTIONS:
Drug: Abemaciclib — twice a day, orally
Drug: Cabozantinib — once daily, orally

SUMMARY:
The researchers are doing this study to find out whether the combination of abemaciclib and cabozantinib is a safe and effective treatment for people with metastatic clear cell renal cell carcinoma (ccRCC) and translocation-associated renal cell cancer (tRCC). The researchers will test different doses of the study drugs to find the highest doses that cause few or mild side effects in participants.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of informed consent
* Patient must be able to provide informed consent, or a legal authorized representative (LAR) must be identified to provide consent in cases where the patient cannot
* Signed and dated IRB-approved Informed Consent Form
* Patient must have a histologically confirmed diagnosis of metastatic stage IV clear cell renal cell carcinoma or metastatic stage IV translocation-associated renal cell carcinoma.
* Patient should have availability of archival tissue that enables definitive diagnosis of ccRCC or tRCC, per review at participating site, accompanied by an associated pathology report. Specimens can be collected by surgical resection or biopsy of the primary tumor or biopsy or resection of a metastatic lesion. NOTE: If archival tissue is unavailable, a patient can still enroll onto the study with documented confirmation from the study PI.
* Patients must have at least one extra-skeletal, extracranial measurable lesion as defined by RECIST v1.1 7. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patients must have progressed on at least 2 prior lines of systemic therapy and a maximum of 3 prior lines of systemic therapy. Prior adjuvant therapy is permitted.
* Patient must have progressed on 1 prior PD-1 or PD-L1 targeted treatment and prior VEGFR directed TKI therapy
* Patients must have recovered to baseline or < Grade 1 CTCAE v5.0 from toxicities related to any prior treatments, unless adverse events (AEs) are clinically non-significant and/or stable on supportive therapy (See Appendix 2)
* Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and registration.
* The patient can swallow oral medications.
* Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment:
* ANC ≥ 1500 cells/μL (without granulocyte colony stimulating factor support within 2 weeks prior to Cycle 1, Day 1)
* WBC counts ≥ 2500/μL and ≤ 15,000/μL without G-CSF
* Absolute Lymphocyte count > 0.5K/mcL
* Platelet count ≥100,000/μL (without transfusion within 2 weeks prior to Cycle 1, Day 1)
* Hemoglobin ≥9.0 g/dL (without transfusion within 2 weeks prior to Cycle 1, Day 1)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 X upper limit of normal (ULN). ALP ≤ 5 x ULN if patient has documented bone metastases.
* Serum bilirubin ≤ 1.5 x ULN. Patients with known Gilbert disease who have serum bilirubin level ≤ 2 x ULN may be enrolled.
* Serum albumin ≥ 2.8 g/dl
* (PT)/INR or partial thromboplastin time (PTT) test < 1.3x the laboratory ULN
* Estimated Glomerular Filtration Rate (eGFR) ≥ 30mL/min using the CKD-EPI formula https://www.kidney.org/professionals/kdoqi/gfr_calculator.
* Urine protein/creatinine ratio (UPCR) ≤ 1.8 mg/mg
* Women of childbearing potential must not be pregnant or lactating at screening.
* Women of childbearing potential who are sexually active with a non-sterilized male partner must use two methods of effective contraception from screening and must agree to continue using such precautions for 4 months after the final dose of investigational product; cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.
* Sexually active participants must agree to use medically accepted methods of contraception (i.e. barrier methods including condoms, female condom, or diaphragm with spermicidal gel) during the study and for 4 months after the last dose of the study treatment. Male patients must agree not to donate sperm during the study treatment period and for 4 months after the last dose Female patients must agree not to donate eggs during the study period and for 4 months after the last dose.

Exclusion Criteria:

* Prior treatment with abemaciclib or cabozantinib.
* Receipt of any type of anti-cancer antibody, cytotoxic anticancer therapy, or any other investigational agents within 2 weeks of treatment start or 5 half-lives, whichever is shorter. For immune checkpoint inhibitors, patients must have discontinued treatment 28 days prior to trial enrollment.
* Symptomatic brain metastasis or leptomeningeal disease requiring steroid use. Patients are eligible if they are neurologically stable for 4 weeks, have completed radiation therapy or surgery, and recovered from side effects. Patients must have discontinued steroid therapy for at least 2 weeks prior to first dose of study treatment.
* Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or early stage cancers previously treated with curative intent.
* Patients requiring moderate or strong CYP3A4 inducers or inhibitors (https://druginteractions.medicine.iu.edu/MainTable.aspx).
* Patients with a history of HIV infection who are not on a stable HAART regimen and/or are requiring antimicrobials for prevention of opportunistic infections and/or have CD4 count below 250 or a detectable HIV viral load
* Patients with active hepatitis B or hepatitis C infection with detectable viral load by PCR
* Active systemic bacterial infection (requiring systemic antibiotics at time of initiating study treatment) or fungal infection.
* History of significant cardiovascular events or active cardiovascular disease; including myocardial infarction within the previous 6 months, unstable arrhythmias, unstable angina, prior sudden cardiac arrest, LVEF < 50% by echocardiogram (ECHO).
* Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
* Significant arterial disease (e.g., stroke, transient ischemic attack, aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Cycle 1, Day 1.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 470 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment.

Note: If a single ECG shows a QTcF with an absolute value > 470 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility

* Concomitant anticoagulation with coumadin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 6 weeks before first dose of study treatment. Completeness of wound healing from any surgery must be ascertained. There must be a minimum of two weeks from completion of wound healing to start of study.
* Evidence of tumor invading the gastrointestinal tract, active peptic ulcer disease, active inflammatory bowel disease, active diverticulitis, active cholecystitis, symptomatic/active cholangitis or appendicitis, acute pancreatitis, acute obstruction of pancreatic duct or common bile duct, or active gastric outlet obstruction.
* Clinical signs or symptoms of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding.
* Patients with a history of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to study enrollment.
* The patient has tumor invading or encasing any major blood vessels, with exception of renal vessels ipsilateral to the primary renal tumor.
* The patient has evidence of tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus) at time of study screening.
* Patients with malabsorption syndrome.
* Patients with a serious non-healing wound/ulcer/bone fracture.
* Patients with active COVID-19 unless the subject has clinically recovered from the disease at least 30 days prior to first dose of study treatment.
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Radiation therapy for bone metastasis within 2 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Maximally Tolerated Dose (MTD) (Phase Ib) | 1 year
  The phase 1b portion of the trial will require between 4 and 24 patients in a 3+3 dose escalation design across four planned separate dose levels. The MTD will be defined as the dose level at which a dose limiting toxicity (DLT) occurs in at most 1 out of 6 patients in that dose level. CTCAE v5.0 will be used for toxicity evaluation.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (Phase II) | 1 year
  per RECIST 1.1 for abemaciclib plus cabozantinib

CONTACTS AND LOCATIONS:
Overall Officials: Martin Voss, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Johns Hopkins University (Data Collection Only), Baltimore, Maryland
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering West Harrison (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm